CLINICAL TRIAL: NCT07012083
Title: Egyptian Doctors' Adherence to Anti-rabies Post-exposure Prophylactic Protocols; A Survey Study
Brief Title: Adherence to Anti-rabies Post-exposure Prophylactic Protocols
Status: Recruiting | Type: Observational
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mohamed Ezzat Nasreddin, Lecturer of Emergency Medicine, Tanta University
Other Study IDs: post exposure anti-rabies
Record Dates: First submitted 2025-05-20; First posted 2025-06-10 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-05

CONDITIONS: Rabies
MeSH Terms: conditions — Rabies | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: survey — This cross-sectional survey study will be conducted on a consecutive sample of physicians who treat patients with animal bites potentially requiring post-exposure anti-rabies prophylaxis. The sample will include emergency physicians, general practice or family physicians, and surgeons of both sexes, with varying degrees of experience and post-graduate clinical training.
  All participants will consent to submit an anonymous Google Form-based questionnaire. The designed questionnaire will include introductory personal, academic, and work experience data about the physicians as gender, age, specialty, workplace, highest achieved medical-academic or training degree, and number of years of postgraduate clinical work experience. Candidates will be asked to reflect on their pre and postgraduate education/training quality and their confidence level in prescribing anti-rabies post-exposure prophylaxis treatment. (as a linear scale).

SUMMARY:
This study aims to investigate physicians' adherence to Advisory Committee on Immunization Practices (ACIP) guidelines regarding Anti-rabies post-exposure prophylaxis in Egypt.

DETAILED DESCRIPTION:
There is no known effective treatment for rabies, and virtually all cases are fatal. Although the prognosis is poor in patients who develop rabies, the disease is usually preventable with proper wound care and post-exposure prophylaxis. Following a thorough risk assessment, the decision to initiate rabies post-exposure prophylaxis should be made. The risk assessment should consider the type of exposure, local rabies epidemiology in animals, vaccination history of the animal, circumstances of the exposure incident, and the availability of the animal for observation or rabies testing .

The World Health Organization (WHO) and the Advisory Committee on Immunization Practices (ACIP) have adopted guidelines for starting post-exposure prophylaxis (PEP) against rabies. The decision to start Anti-Rabies PEP is usually made in primary health care units or emergency departments .

Lack of adherence to these guidelines might result in unnecessary costs and medical risks, such as injection site reactions and systemic hypersensitivity reactions . This malpractice of inappropriate anti-rabies PEP prescription is not uncommon.

ELIGIBILITY:
Inclusion Criteria:

* Physicians who treat patients with animal bites potentially requiring post-exposure anti-rabies prophylaxis. The sample will include emergency physicians, general practice or family physicians, and surgeons of both sexes, with varying degrees of experience and post-graduate clinical training.

Exclusion Criteria:

* Incomplete record filling

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This cross-sectional survey study will be conducted on a consecutive sample of physicians who treat patients with animal bites potentially requiring post-exposure anti-rabies prophylaxis. The sample will include emergency physicians, general practice or family physicians, and surgeons of both sexes, with varying degrees of experience and post-graduate clinical training.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Adherence to Anti-rabies PEP Guidelines | 6 months
  This study aims to investigate physicians' adherence to the Advisory Committee on Immunization.
  Practices (ACIP) guidelines regarding Anti-rabies post-exposure prophylaxis in Egypt. This will be through a score given for the correct response to the case-based questionnaire. This questionnaire include 10 case-based scenarios where anti-rabies post-exposure prophylaxis may or may not be indicated as per ACIP guidelines. True response will be scored 1, wrong response will be scored 0 with maximum total score of 10. Higher score reflects better adherence to guidelines recommendations & vice versa.

SECONDARY OUTCOMES:
Health & Economic burden of such malpractice | 9 months
  This study attempts to evaluate the possible economic burden of this expected departure from the standard of care by examining doctors' compliance with appropriate prescription of anti-rabies post-exposure prophylaxis. Economic burden will be calculated by incorporating total odds ratio of inappropriate prescription of anti-rabies vaccine with or without human rabies immunoglobulin , cost of each dose of them to get a rough estimate of the expected cost rising from inappropriate prescription of theses drugs when they are not indicated.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine Tanta university, Tanta, Gharbia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Catherine M Brown, Alfred DeMaria. Indications for post-exposure rabies prophylaxis In: UpToDate, Connor RF (Ed), Wolters Kluwer. (Accessed on Oct 15, 2024).
- [Background] Protocol for a well-performed rabies post-exposure prophylaxis delivery: To read along with the decision trees, 1- Wound Risk Assessment and 2 - PEP Risk Assessment. Geneva: World Health Organization; 2024. https://doi.org/10.2471/ B09018.
- [Background] Rupprecht CE, Briggs D, Brown CM, Franka R, Katz SL, Kerr HD, Lett SM, Levis R, Meltzer MI, Schaffner W, Cieslak PR; Centers for Disease Control and Prevention (CDC). Use of a reduced (4-dose) vaccine schedule for postexposure prophylaxis to prevent human rabies: recommendations of the advisory committee on immunization practices. MMWR Recomm Rep. 2010 Mar 19;59(RR-2):1-9. PMID 20300058